CLINICAL TRIAL: NCT05440786
Title: A Randomized, Open-Label, Phase 2 Study Evaluating Abemaciclib in Combination With Irinotecan and Temozolomide in Participants With Relapsed or Refractory Ewing's Sarcoma
Brief Title: CAMPFIRE: A Study of Abemaciclib (LY2835219) in Participants With Ewing's Sarcoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18434; J1S-MC-JP04 (Other: Eli Lilly and Company); 2023-506772-28-00 (EU CTIS Number)
Expanded Access: NCT03763604 (Approved for marketing)
Record Dates: First submitted 2022-06-28; First posted 2022-07-01 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Sarcoma, Ewing; Neoplasm Metastasis
MeSH Terms: conditions — Sarcoma, Ewing; Neoplasm Metastasis | interventions — abemaciclib; Irinotecan; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Abemaciclib + Irinotecan +Temozolomide (Experimental): Abemaciclib given orally in combination with irinotecan given IV and temozolomide given orally.
  Interventions: Drug: Abemaciclib; Drug: Irinotecan; Drug: Temozolomide
- Irinotecan +Temozolomide (Experimental): Irinotecan given IV and temozolomide orally.
  Interventions: Drug: Irinotecan; Drug: Temozolomide

INTERVENTIONS:
Drug: Abemaciclib — Orally
  Other Names: LY2835219
  Arms: Abemaciclib + Irinotecan +Temozolomide
Drug: Irinotecan — IV
Drug: Temozolomide — Orally

SUMMARY:
The purpose of this study is to measure the benefit of adding abemaciclib to chemotherapy (irinotecan and temozolamide) for Ewing's sarcoma that has come back or did not respond to treatment. This trial is part of the CAMPFIRE master protocol, which is a platform to speed development of new treatments for children and young adults with cancer. Your participation in this trial could last 11 months or longer, depending on how you and your tumor respond.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Ewing's sarcoma or Ewing's sarcoma-like tumor by institutional pathologist. The original pathological report is required. Repeat biopsy at progression is not required
* Refractory disease or confirmed radiological progression or recurrence following first or later line of treatment of Ewing's sarcoma or Ewing's sarcoma-like tumor

  -- Must have one measurable or evaluable lesion per RECIST 1.1
* Adequate performance status based on age

  * For participants less than (<)16 years of age, a Lansky score greater than or equal to (≥)50, or
  * For participants ≥16 years of age, a Karnofsky score ≥50
* Participants must have discontinued all previous treatments for cancer or investigational agents ≥7 days after the last dose and must have recovered from the acute effects
* Adequate hematologic and organ function less than or equal to (≤)14 days prior to Day 1 of Cycle 1:

  * Absolute neutrophil count ≥1000/microliter (µL)
  * Platelets ≥75,000/cubic millimeter (mm³)
  * Hemoglobin ≥8 grams per deciLiter (g/Dl) (≥100 grams per Liter [g/L])
  * Total bilirubin ≤1.5 times (×) upper limit of normal (ULN)
  * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤3 × ULN
  * Creatinine clearance or calculated glomerular filtration rate (GFR) ≥60 milliliters per minute per square meter (Ml/min/m²) or serum creatinine based on age/gender
* Female participants of childbearing potential must have a negative urine or serum pregnancy test
* Body weight ≥10 kilograms (kg)
* Must be able to swallow and/or have a gastric/nasogastric tube

  -- Participants in the European Union must be able to swallow intact capsules
* Stable or decreasing dose of steroids at least 7 days prior to enrollment
* Life expectancy of at least 8 weeks and able to complete at least 1 cycle of treatment
* Participants/caregivers are able and willing to make themselves available for the duration of the study and are willing to follow study procedures, including adherence to the pharmacokinetic (PK) sampling schedule

Exclusion Criteria:

* Participants with severe and/or uncontrolled concurrent medical disease or psychiatric illness/social situation that in the opinion of the investigator could cause unacceptable safety risks or compromise compliance with the protocol
* Participants with an active fungal, bacterial, and/or known severe viral infection including, but not limited to, human immunodeficiency virus (HIV) or viral (A, B, or C) hepatitis.
* Participants who have had allogeneic bone marrow or solid organ transplant
* Surgery: Participants who have had, or are planning to have, the following invasive procedures:

  * Major surgical procedure, laparoscopic procedure, or significant traumatic injury within 28 days prior to enrollment
  * Surgical or other wounds must be adequately healed prior to enrollment
* Female participants who are pregnant or breastfeeding
* Have received any prior cyclin-dependent kinase (CDK) 4 and 6 inhibitor
* Progression during prior treatment with irinotecan and/or temozolomide
* Have a known intolerability or hypersensitivity to any of the study treatments or dacarbazine
* Diagnosed and/or treated additional malignancy within 3 years prior to enrollment

Ages: 1 Year to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 45 (Estimated)
Dates: Start 2022-09-20 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | Baseline to objective progression or death due to any cause (estimated up to 11 months)
  PFS determined by blinded independent review committee (BIRC) using Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST 1.1)

SECONDARY OUTCOMES:
Overall Survival (OS) | Baseline to date of death due to any cause (estimated up to 45 months)
  OS
Overall Response Rate (ORR): Percentage of Participants Who Achieve Complete Response (CR) or Partial Response (PR | Baseline to measured progressive disease (estimated up to 11 months)
  ORR
Duration of Response (DoR) | Date of first evidence of CR or PR to date of disease recurrence, objective disease progression, or death due to any cause (estimated up to 11 months)
  DoR
Disease Control Rate (DCR) | Baseline to measured progressive disease (estimated up to 11 months)
  DCR
PFS | Baseline to objective progression or death due to any cause (estimated up to 11 months)
  PFS determined by investigator assessment using RECIST 1.1
Pharmacokinetics (PK): Minimum Plasma Concentration (Cmin) of Abemaciclib | Cycle 3, Day 1 (21 day cycles)
  PK: Cmin of Abemaciclib
Abemaciclib Product Acceptability | Day 1 of Cycles 1 through 3 (21 day cycles)
  Participants evaluated abemaciclib acceptability (palatability and ease of administration) using a 5-category questionnaire. Participants were asked to select one of the following to describe the acceptability of abemaciclib: Very difficult, difficult, neither easy nor difficult, easy, or very easy.

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (28):
- United States (5):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - The Regents of the University of California - Los Angeles (UCLA Pediatrics), Los Angeles, California
  - Riley Hospital for Children at Indiana University Health, Indianapolis, Indiana
  - Washington University, St Louis, Missouri
  - Lifespan Cancer Institute, Providence, Rhode Island
- Australia (3):
  - The Children's Hospital at Westmead, Westmead, New South Wales
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - Royal Children's Hospital, Melbourne, Victoria
- France (2):
  - Institut Bergonié - Centre Régional de Lutte Contre Le Cancer de Bordeaux et Sud Ouest, Bordeaux, Aquitaine
  - Centre Leon Berard, Lyon, Auvergne-Rhône-Alpes
- Germany (3):
  - Universitaetsklinikum Freiburg, Freiburg im Breisgau, Baden-Wurttemberg
  - Universitätsklinikum Essen, Essen, North Rhine-Westphalia
  - Charité Campus Virchow-Klinikum, Berlin
- Italy (2):
  - Fondazione Policlinico Universitario Agostino Gemelli, Rome, Lazio
  - IRCCS Istituto Ortopedico Rizzoli, Bologna
- Japan (3):
  - Hyogo Prefectural Kobe Children's Hospital, Kobe, Hyōgo
  - National Cancer Center Hospital, Chuo-ku, Tokyo
  - Kyushu University Hospital, Fukuoka
- Spain (10):
  - Hospital Universitari Vall d'Hebron, Barcelona, Barcelona [Barcelona]
  - Hospital Sant Joan de Déu, Esplugues de Llobregat, Barcelona [Barcelona]
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Catalunya [Cataluña]
  - Hospital Infantil Universitario Niño Jesús, Madrid, Madrid, Comunidad de
  - Hospital Universitario La Paz, Madrid, Madrid, Comunidad de
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Virgen Del Rocio, Seville
  - Hospital Universitari i Politecnic La Fe, Valencia

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/

REFERENCES:
- See also: CAMPFIRE: A Study of Abemaciclib (LY2835219) in Participants With Ewing's Sarcoma — https://trials.lillytrialguide.com/en-US/trial/6ZWD0uc8v7H8M6hyLyDv9e